CLINICAL TRIAL: NCT03717662
Title: Promoting Women's Health: A Gender Specific Smoking Cessation Program for Female Smokers in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 06-323
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Smoking Cessation
Keywords: women
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief counseling and NRT (Experimental): The project will provide intensive counseling at the Centre for Health Promotion (CHP) of HKU Department of Nursing Studies, female smokers (including all types of tobacco products such as shisha, electronic cigarettes and heat-not-burn (HNB) which are available in the market) who require more intensive counseling or advice on nicotine replacement therapy, upon referral from the women's organizations and trained women counselors. The smokers will receive face-to-face (or telephone) counseling and a 1 week supply of Nicotine replacement therapy (NRT) (4 mg nicotine gum or 10 mg/ 15 mg nicotine patch) from the nurse counselor, and follow up calls at 1 week, 1-, 3-, 6-, 36- and 72-month post-intervention.
  Interventions: Drug: nicotine gum or nicotine patch

INTERVENTIONS:
Drug: nicotine gum or nicotine patch — The project will provide intensive counseling at the Centre for Health Promotion (CHP) of HKU Department of Nursing Studies, female smokers who require more intensive counseling or advice on nicotine replacement therapy, upon referral from the women's organizations and trained women counselors. The smokers will receive face-to-face (or telephone) counseling and a 1 week supply of Nicotine replacement therapy (NRT) (4 mg nicotine gum or 10 mg/ 15 mg nicotine patch) from the nurse counselor, and follow up calls at 1 week, 1-, 3-, 6-, 36- and 72-month post-intervention.

SUMMARY:
This project aims to publicize quitting among female smokers, and encourage and support those who want to quit by providing face-to-face and/or telephone counseling. The objectives are to:

1. Build up a Women Against Tobacco Taskforce (WATT) with woman volunteers from various organizations to promote quitting in female smokers, and to arouse public awareness of the effects of smoking on sexual, reproductive and child health, and other diseases among women.
2. Conduct a survey among the women volunteers and staff of the women's organization to ascertain their learning needs, knowledge, attitudes, and practice of tobacco control and smoking cessation, and to identify interested participants to join the smoking cessation training program.
3. Design and deliver a smoking cessation counseling training program (based on the learning needs identified), to equip women volunteers with the knowledge and skills in smoking cessation.
4. Develop and evaluate a gender-specific smoking cessation program to help female smokers to reduce and quit smoking.
5. Promote women's health and quality of life, and reduce the life-long morbidity and mortality of female smokers in the long term.
6. Examine the long term (3-year) impact of a gender-specific smoking cessation program on the smoking behaviors of female smokers.
7. Examine another long-term (6-year) impact of a gender-specific smoking cessation program on the smoking behaviors of female smokers.
8. Ascertain the contributing factors in the rate of quitting, retention and relapse.
9. Investigate Hong Kong women smokers awareness and attitude to women quitline.

DETAILED DESCRIPTION:
Phase I: Build up a network and need assessment

1. We will invite collaboration with the Hong Kong Women Development Association (18 organizational members and over 30,000 individual members), the Hong Kong Federation of Women (45 organizational members), Women's Club of Family Planning Association (7 Women's Club), Hone Kong Young Women's Christian Association (around 260,000 members) and other woman organizations to build up a network by setting up a Women Against Tobacco Taskforce (WATT) jointly with representatives from women organizations and led by the Department of Nursing Studies of The University of Hong Kong. This proposed Task Force will focus on promoting smoking cessation among female smokers and arousing the public's awareness of health risks specific to women from smoking.
2. Need assessment survey and focus group interview of the women volunteers and staff: all volunteers and staff will be invited to participate in a need assessment survey and focus group interview. The perceived needs identified will be used to design a tailor-made smoking cessation counselor training curriculum for the participants, and they will be asked to indicate their interest and commitment to undertake such training (free of charge), and to help women quit smoking.

Phase II:

Design and deliver training curriculum: Based on the needs assessment data, we will design and deliver a tailor-made smoking cessation counseling training program for the woman volunteers and staff. A maximum capacity of 200 participants can be trained. At the end of the program, participants should be capable of delivering smoking cessation advice for women, and a referral system can be set up so that women that required more intensive counseling can be referred to us if necessary. The outcome of the training will be evaluated through a survey before and immediate after, and 6 months post training, which include: knowledge, attitudes, and practice of smoking cessation.

We aim to train women smoking cessation counselors as they can better understand the needs and feelings of female smokers. Female addiction to cigarette smoking may be reinforced more by the sensory and social context of smoking2, and therefore it is important to reduce the gap between the female smoker and the counselor. Upon completion of the program, a certificate of attendance will be awarded to the participants and their organizations for their contribution.

Phase III:

1. Brief gender-specific advice provided by trained women volunteers: The trained women counselors will use motivational approach to provide smoking cessation advice to female smokers.
2. Intensive gender-specific intervention provided by experience nurse counselor: The project will provide intensive counseling at the Centre for Health Promotion (CHP) of HKU Department of Nursing Studies, female smokers (including all types of tobacco products such as shisha, electronic cigarettes and heat-not-burn (HNB) which are available in the market) who require more intensive counseling or advice on nicotine replacement therapy, upon referral from the women's organizations and trained women counselors. The smokers will receive face-to-face (or telephone) counseling and a 1 week supply of Nicotine replacement therapy (NRT) (4 mg nicotine gum or 10 mg/ 15 mg nicotine patch) from the nurse counselor, and follow up calls at 1 week, 1-, 3-, 6-, 36- and 72-month post-intervention. Their smoking status, information about usage of nicotine replacement products and quality of life measures will be assessed. All women reported to have quit smoking at 6-, 36- and 72-month will be invited for biochemical validation (measurement of urine / saliva cotinine level). Participants will be invited to do qualitative interviews (individual / focus group interviews) at the 36-month follow up. Interviews will be conducted according to participants' smoking status (3 levels: continuous smoker; those who had quit attempts but relapsed; and those who abstained from tobacco within the 3-year period) and martial status (2 levels: single; and married). 30 participants with 5 subjects per group will be recruited. Each interview will last for 60 minutes and to be conducted by an experienced facilitator at the School of Nursing, The University of Hong Kong. During each individual interview, the facilitator will first welcome the participants, obtain written consent, and assure that the interview will be audio-taped and kept confidential. The facilitator will guide the discussion using an interview guide and prompt for further information as necessary.

Phase IV:

The trained women counsellors will observe the women smokers on the street and walk forward to look for opportunities talking to them. Counsellors will first explain the basic information of this research and acquire their reliance. After we got the permission to conduct a small interview, smokers will be asked a few questions about their awareness about women quitline and obstruction to call the quitline. Each interview will last no more than 10 minutes. We can invite them to participate in a further phone call survey and encourage them to leave their phone number.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong female resident aged 18 or above
* Able to communicate in Chinese (Cantonese)
* Current Smokers

Exclusion Criteria:

* Have difficulty to communicate via telephone
* Having queries irrelevant to tobacco control

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only female smokers will be selected.
Enrollment: 480 (Estimated)
Dates: Start 2006-04-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
7-days point prevalence smoking abstinence at 6-month | 6-month follow-up
  the reduced cigarette consumption; progression to a higher stage of readiness to change; quit attempts, and increased self-efficacy to quitting smoking. In the long term, the quit rate (not smoke for at least 7 days during the time of follow up); smoking reduction, progression of stage of readiness, at 6 months; and change in quality of life

SECONDARY OUTCOMES:
Bio-chemical validated smoking abstinence at 6-,36-,72-month | 6-,36-,72-month follow-up
  Bio-chemical validated smoking abstinence is measured at 6-,36-,72-month. The participants who claim to have quitted smoking for at least 7 days are invited for biochemical validation (measurement of saliva cotinine level and exhaled carbon monoxide level) at 6-month. The participants are need to get the results of CO≤ 4ppm, and continine level ≤30 ng/ml as passing results.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Cheung Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No